CLINICAL TRIAL: NCT02648646
Title: Falls Prevention Program for Adults With Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-1448
Record Dates: First submitted 2015-11-02; First posted 2016-01-07 (Estimated); Results first posted 2018-10-26 (Actual); Last update posted 2018-10-26 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis; Falls, Accidental
MeSH Terms: conditions — Osteoarthritis | interventions — Walking; methyl hydroxyethyl cellulose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm - Intervention (Experimental): Receives Otago Exercise Programme and Walk with Ease
  Interventions: Other: Otago Exercise Programme and Walk with Ease

INTERVENTIONS:
Other: Otago Exercise Programme and Walk with Ease — The Otago Exercise Programme is a falls prevention program that is successful at reducing falls in adults 65+ years of age. Briefly, this program includes flexibility, progressive lower extremity strengthening with ankle weights, and balance exercises. The investigators are replacing the Otago walking program with the evidence-based Arthritis Foundation's Walk With Ease program.

SUMMARY:
Purpose: To report the feasibility and to obtain preliminary data on the effects of using an enhanced Otago Exercise Programme to reduce fall risk in individuals with osteoarthritis (OA).

Participants: Ten participants from the Johnston County Osteoarthritis Project who have OA, are at risk for falls, and are 65+ years old.

Procedures (methods): All participants will receive the 6-month enhanced Otago program. The investigators will assemble data: quantifying participant adherence to and safety of the intervention, ascertaining retention of participants for 6 months, determining acceptability of the program, and other validated measures (e.g., number of falls and fall severity, balance measures).

ELIGIBILITY:
Inclusion Criteria:

* history of falls
* knee or hip radiographic OA
* 65+ years of age
* normal cognitive function (based on the Mini-Mental State Examination)
* current knee/hip symptoms

Exclusion Criteria:

* hospitalized for stroke, myocardial infarction, or coronary artery revascularization in past 3 months
* diagnosis of metastatic cancer in the past 3 months
* terminal illness
* progressive neurological disorders
* rheumatoid arthritis
* severe fibromyalgia
* other systemic rheumatic disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-11-02 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Golightly, PT, PhD, Principal Investigator — University of North Carolina, Chapel Hill

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Arm - Intervention
Started | 10
Completed | 8
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 10
Age, Continuous [Median (Full Range); unit: years] | 71.3 [65.4 to 79.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Participant Adherence to Intervention
Description: Number of participants who adhere to the intervention.
Time Frame: 6 months
Population: 8 participants completed the 6-month intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
Participants | 5

2. Primary Outcome: Participant Safety With the Intervention
Description: Number and type of adverse events related to the intervention.
Time Frame: 6 months
Population: 8 participants completed the 6-month intervention
Measure: Number; unit: adverse events
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
adverse events | 0

3. Primary Outcome: Retention of Participants
Description: Number of participants who participate in the study for the full 6 month program.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 10
Participants
  Completed | 8
  Reason not completed: total knee replacement | 1
  Reason not compelted: Injury not related to study | 1

4. Primary Outcome: Acceptability of the Program
Description: Descriptive summary of participants' reports from closing interview of what they like and do not like about the program, any challenges they experienced with doing the program, and whether they plan to continue what they learned.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
Participants
  Liked exercising with this program | 2
  The program helped individual move better | 3
  Exercises were easy | 1
  Liked the program gave structure | 1
  Liked that program promoted working towards goals | 1
  Did not like Walk With Ease workbook, hard to use | 1
  One exercise hurt hip; PT changed it & was fin | 1
  Reported no dislikes of program | 6
  Challenge of program: standing on 1 foot | 3
  Challenge of program: needed to hold onto counter | 1
  Exercises were challenging at first | 1
  Challenging to learn new exercises | 1
  Challenge to make self do program on own | 1
  No challenges with program | 1
  Plans to continue to practice what they learned | 8

5. Secondary Outcome: Number of Falls
Description: Participant will record occurrence of falls on a monthly falls calendar. Number of falls over the 6 month program will be calculated.
Time Frame: Baseline to Month 6
Measure: Number; unit: falls
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
falls | 3

6. Secondary Outcome: Number of People With Severe of Falls
Description: Participant will record whether the fall resulted in an injury and the type of injury that occurred. A fall will be considered severe if an injury occurred.
Time Frame: Baseline to Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
Participants | 1

7. Secondary Outcome: Berg Balance Scale
Description: This is 14 item scale that measures balance among older adults. The participant attempts to complete 14 different balance tests (e.g., stand unsupported with eyes closed, pick up object from floor from standing position), closely supervised by a physical therapist to prevent fall or injury. The test takes no more than 15 minutes to complete and a total score is calculated of 0-56 (high fall risk to low fall risk).
Time Frame: Baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 47.5 [39 to 52]

8. Secondary Outcome: Four-tests Balance: Feet Together Stand
Description: Four timed static balance tasks of increasing difficulty are completed without assistive devices: 1) feet together stand for up to 10 seconds; 2) semi-tandem stand (heel of one foot placed to the side of the big toe of the other foot) for up to 10 seconds; 3) tandem stand (one foot in front of the other, heel touching toe) for up to 10 seconds; and 4) one leg stand for up to 30 seconds. Time for each test is recorded in seconds. If the participant cannot achieve a task, this is recorded as 0 seconds.
Time Frame: Baseline
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 10 [0 to 10]

9. Secondary Outcome: Hand Grip Dynamometry Right Hand
Description: Participant squeezes hand dynamometer with maximum strength, and force is recorded in kgs.
Time Frame: Baseline
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
kilograms | 15.7 [9.3 to 26.7]

10. Secondary Outcome: 30-second Chair Stand Test
Description: Participant rises from chair to full standing position and sits back down as quickly as possible for 30 seconds. Number of completed sit to stand to sit maneuvers is recorded.
Time Frame: Baseline
Measure: Median (Full Range); unit: completed maneuvers
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
completed maneuvers | 9 [6 to 14]

11. Secondary Outcome: Timed Up and Go Test
Description: Participant stands up from chair, walks 3 meters, turns around, walks back to chair, and sits down. Time to complete task is recorded in seconds.
Time Frame: Baseline
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 21.6 [12.2 to 27.3]

12. Secondary Outcome: Stair Climb Test
Description: Participant ascends and descends 3 stairs as quickly as possible in a safe manner, using handrail and walking aid if needed. Time to complete task is recorded in seconds.
Time Frame: Baseline
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 9.8 [6.5 to 15.9]

13. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index
Description: This questionnaire include 5 questions about knee or hip pain, 2 questions about knee or hip stiffness, and 17 questions about difficulty with performing daily activities that involve the lower body. Each item is scored from 0-4 (none, slight, moderate, severe, and extreme). A total score is calculated by summing the item scores and ranges from 0 (no problems) to 96 (extreme problems).
Time Frame: Baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 37 [15 to 46]

14. Secondary Outcome: Activities-specific Balance Confidence Scale
Description: Participant reports level of confidence in doing an activity without losing balance or becoming unsteady on a scale of 0-100%. The ratings are totaled and divided by 16 (the number of items) to calculate a total score.
Time Frame: Baseline
Measure: Median (Full Range); unit: percentage of confidence
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
percentage of confidence | 64.1 [25.0 to 78.8]

15. Secondary Outcome: Rapid Assessment of Physical Activity: Aerobic Score
Description: Participants are asked to identify from a list of 7 items which one accurately describes their current level of aerobic physical activity. Participants who identify with items 6 or 7 are considered active. Those who identify with items 1-5 are considered to have suboptimal aerobic physical activity levels.
  Sedentary:
  1. I rarely or never do any physical activities.
     Under-active:
  2. I do some light or moderate physical activities, but not every week.
     Under-active regular - light activities:
  3. I do some light physical activity every week.
     Under-active regular:
  4. I do moderate physical activities every week, but less than 30 minutes a day or 5 days a week.
  5. I do vigorous physical activities every week, but less than 20 minutes a day or 3 days a week.
     Active:
  6. I do 30 minutes or more a day of moderate physical activities, 5 or more days a week.
  7. I do 20 minutes or more a day of vigorous physical activities, 3 or more days a week.
Time Frame: Baseline
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 3.5 [2 to 7]

16. Secondary Outcome: Berg Balance Scale
Description: as for outcome 7
Time Frame: Week 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 49.5 [44 to 53]

17. Secondary Outcome: Berg Balance Scale
Description: as for outcome 7
Time Frame: Month 6
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 48 [43 to 56]

18. Secondary Outcome: Four-tests Balance: Feet Together Stand
Description: as for outcome 8
Time Frame: Week 8
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 10.0 [2.3 to 10.0]

19. Secondary Outcome: Four-tests Balance: Feet Together Stand
Description: as for outcome 8
Time Frame: Month 6
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 10.0 [10.0 to 10.0]

20. Secondary Outcome: Four-tests Balance: Semi-tandem Stand
Description: as for outcome 8
Time Frame: Baseline
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 10.0 [0.0 to 10.0]

21. Secondary Outcome: Four-tests Balance: Semi-tandem Stand
Description: as for outcome 8
Time Frame: Week 8
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 7.4 [0.0 to 10.0]

22. Secondary Outcome: Four-tests Balance: Semi-tandem Stand
Description: as for outcome 8
Time Frame: Month 6
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 10.0 [10.0 to 10.0]

23. Secondary Outcome: Four-tests Balance: Tandem Stand
Description: as for outcome 8
Time Frame: Baseline
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 10.0 [0.0 to 10.0]

24. Secondary Outcome: Four-tests Balance: Tandem Stand
Description: as for outcome 8
Time Frame: Week 8
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 0.0 [0.0 to 10.0]

25. Secondary Outcome: Four-tests Balance: Tandem Stand
Description: as for outcome 8
Time Frame: Month 6
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 5.2 [0.0 to 10.0]

26. Secondary Outcome: Four-tests Balance: One Leg Stand
Description: as for outcome 8
Time Frame: Baseline
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 0.0 [0.0 to 9.0]

27. Secondary Outcome: Four-tests Balance: One Leg Stand
Description: as for outcome 8
Time Frame: Week 8
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 0.0 [0.0 to 10.0]

28. Secondary Outcome: Four-tests Balance: One Leg Stand
Description: as for outcome 8
Time Frame: Month 6
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 0.9 [0.0 to 28.0]

29. Secondary Outcome: Hand Grip Dynamometry Right Hand
Description: Participant squeezes hand dynamometer with maximum strength, and force is recorded in kgs.
Time Frame: Week 8
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
kilograms | 15.0 [10.7 to 28.0]

30. Secondary Outcome: Hand Grip Dynamometry Right Hand
Description: Participant squeezes hand dynamometer with maximum strength, and force is recorded in kgs.
Time Frame: Month 6
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
kilograms | 17.7 [14.7 to 24.7]

31. Secondary Outcome: Hand Grip Dynamometry Left Hand
Description: Participant squeezes hand dynamometer with maximum strength, and force is recorded in kgs.
Time Frame: Baseline
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
kilograms | 17.0 [10.7 to 24.0]

32. Secondary Outcome: Hand Grip Dynamometry Left Hand
Description: Participant squeezes hand dynamometer with maximum strength, and force is recorded in kgs.
Time Frame: Week 8
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
kilograms | 16.7 [7.3 to 26.7]

33. Secondary Outcome: Hand Grip Dynamometry Left Hand
Description: Participant squeezes hand dynamometer with maximum strength, and force is recorded in kgs.
Time Frame: Month 6
Measure: Median (Full Range); unit: kilograms
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
kilograms | 16.7 [10.0 to 24.7]

34. Secondary Outcome: 30-second Chair Stand Test
Description: as for outcome 10
Time Frame: Week 8
Measure: Median (Full Range); unit: completed maneuvers
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
completed maneuvers | 7.5 [6 to 16]

35. Secondary Outcome: 30-second Chair Stand Test
Description: as for outcome 10
Time Frame: Month 6
Measure: Median (Full Range); unit: completed maneuvers
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
completed maneuvers | 9 [8 to 20]

36. Secondary Outcome: Timed Up and Go Test
Description: as for outcome 11
Time Frame: Week 8
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 19.5 [14.5 to 28.8]

37. Secondary Outcome: Timed Up and Go Test
Description: as for outcome 11
Time Frame: Month 6
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 16.8 [14.5 to 29.5]

38. Secondary Outcome: Stair Climb Test
Description: as for outcome 12
Time Frame: Week 8
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 9.0 [7.1 to 17.5]

39. Secondary Outcome: Stair Climb Test
Description: as for outcome 12
Time Frame: Month 6
Measure: Median (Full Range); unit: seconds
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
seconds | 8.8 [5.3 to 16.9]

40. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index
Description: as for outcome 13
Time Frame: Week 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 7
units on a scale | 31 [9 to 52]

41. Secondary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index
Description: as for outcome 13
Time Frame: Month 6
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 23.5 [16 to 41]

42. Secondary Outcome: Activities-specific Balance Confidence Scale
Description: as for outcome 14
Time Frame: Week 8
Measure: Median (Full Range); unit: percentage of confidence
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
percentage of confidence | 60.6 [51.9 to 80.6]

43. Secondary Outcome: Activities-specific Balance Confidence Scale
Description: as for outcome 14
Time Frame: Month 6
Measure: Median (Full Range); unit: percentage of confidence
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
percentage of confidence | 59.1 [31.3 to 81.3]

44. Secondary Outcome: Rapid Assessment of Physical Activity: Aerobic Score
Description: as for outcome 15
Time Frame: Week 8
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 4 [3 to 7]

45. Secondary Outcome: Rapid Assessment of Physical Activity: Aerobic Score
Description: as for outcome 15
Time Frame: Month 6
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Single Arm - Intervention
Number analyzed (Participants) | 8
units on a scale | 4 [3 to 6]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Single Arm - Intervention
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm - Intervention (N=10)
Fall (Injury, poisoning and procedural complications) | 1 (1) — One participant fell while walking quickly in flip-flop shoes in her apartment parking lot during Month 5. She injured her elbow (requiring 8 stitches from the urgent care) and bruised her knee, but was recovering well by Month 6 visit.
Fall (Injury, poisoning and procedural complications) | 1 (1) — Participant fell during Month 4 when she got up to go to bathroom during the middle of the night. Her blood pressure dropped and she felt faint; she slid slowly to the floor but was not injured.
Fall (Injury, poisoning and procedural complications) | 1 (1) — The participant fell during Month 4 when she tripped over a vine in her yard. She was not injured.
Injury (Injury, poisoning and procedural complications) | 1 (1) — The participant injured his hips lifting a wheelchair prior to the Week 4 visit and withdrew from the study because of this injury (which was not related to the study).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No